CLINICAL TRIAL: NCT07265388
Title: Validation and Extension of the SUCCESS Score for Fuchs Dystrophy After Cataract Surgery
Brief Title: SUCCESS Score Validation in Fuchs Dystrophy
Acronym: SUCCESS
Status: Recruiting | Type: Observational
Sponsor: Instituto Ramón y Cajal de Investigación Sanitaria (Other)
Responsible Party: Principal Investigator, Francisco Arnalich-Montiel, Lead investigator of the Ophtalmology department, Instituto Ramón y Cajal de Investigación Sanitaria
Other Study IDs: SUCCESS-FUCHS; PI22/01252 (Other Grant/Funding Number: Instituto de Salud Carlos III (ISCIII))
Record Dates: First submitted 2025-11-24; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Fuchs Endothelial Corneal Dystrophy
Keywords: Fuchs Endothelial Corneal Dystrophy; Cataract Surgery; endothelial keratoplasty; Diagnostic Accuracy; Prognostic Validation; Predictive Modeling
MeSH Terms: conditions — Fuchs' Endothelial Dystrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- FECD Cohort: Patients with clinically diagnosed Fuchs endothelial corneal dystrophy (FECD) undergoing phacoemulsification cataract surgery at participating tertiary centers. All participants receive standard cataract surgery, and their preoperative data are used to calculate the SUCCESS Score with and without corneal densitometry parameters. Postoperative outcomes are monitored to determine the need for endothelial keratoplasty (EK).
  Interventions: Procedure: Phacoemulsification Cataract Surgery

INTERVENTIONS:
Procedure: Phacoemulsification Cataract Surgery — Standard phacoemulsification cataract surgery performed in patients with Fuchs endothelial corneal dystrophy (FECD). All procedures are carried out according to institutional protocols at participating tertiary centers. Preoperative Scheimpflug tomography and corneal densitometry measurements are collected to calculate the SUCCESS Score and evaluate the risk of postoperative endothelial decompensation. Postoperative outcomes are monitored to determine whether endothelial keratoplasty (EK) is required during follow-up.

SUMMARY:
This prospective multicenter diagnostic study aims to externally validate and extend the SUCCESS Score for predicting the need for endothelial keratoplasty after cataract surgery in patients with Fuchs endothelial corneal dystrophy (FECD). The model's performance and clinical utility are assessed using discrimination, calibration, and reclassification metrics.

DETAILED DESCRIPTION:
Fuchs endothelial corneal dystrophy (FECD) is a progressive corneal disorder characterized by endothelial cell loss, corneal edema, and visual impairment. In patients with FECD and cataract, an important clinical challenge is to predict whether cataract surgery alone will suffice or whether endothelial keratoplasty (EK) will be required postoperatively. Accurate preoperative risk stratification is essential for surgical planning and patient counseling.

The SUCCESS Score, derived from Scheimpflug tomography, was proposed as an objective index to estimate the risk of postoperative corneal decompensation in FECD. However, its external multicenter validation and the potential contribution of corneal densitometry have not yet been fully established.

This ongoing prospective, observational, multicenter study aims to externally validate and extend the SUCCESS Score for predicting the need for EK after cataract surgery in patients with FECD. The study is being conducted across five tertiary referral centers in Spain. Eligible participants are adults with FECD grade ≥2 on the modified Krachmer scale and a visually significant cataract requiring phacoemulsification. Patients with epithelial edema, prior ocular surgery, corneal infection, or trauma are excluded.

Preoperative evaluation includes Scheimpflug tomography and corneal densitometry analysis. The primary outcome is the requirement for endothelial keratoplasty after cataract surgery, determined by postoperative visual function and corneal evaluation. Model performance will be assessed through discrimination (Harrell's C statistic), calibration, reclassification (IDI, NRI), and decision curve analysis to estimate clinical utility.

The primary analysis is scheduled for completion in October 2024. Extended follow-up will continue until June 25, 2026, to assess long-term predictive performance and generalizability of the extended SUCCESS model.

An interactive web-based calculator implementing both the original and extended SUCCESS models will be provided as a supplementary tool to facilitate clinical use and standardized patient counseling across participating centers.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥40 years.
* Clinical diagnosis of Fuchs endothelial corneal dystrophy (FECD) grade ≥2 on the modified Krachmer scale.
* Presence of visually significant cataract requiring phacoemulsification surgery.
* Ability to provide informed consent and comply with study procedures.
* Availability of preoperative Scheimpflug tomography and corneal densitometry measurements.

Exclusion Criteria:

* Epithelial or stromal edema precluding reliable corneal imaging.
* Previous ocular surgery (including corneal or intraocular procedures).
* Corneal trauma, infection, or inflammation affecting endothelial integrity.
* Coexisting ocular pathologies that could confound postoperative assessment (e.g., advanced glaucoma, macular degeneration).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: dults with clinically diagnosed Fuchs endothelial corneal dystrophy (FECD) and visually significant cataract who are scheduled to undergo phacoemulsification surgery at participating tertiary referral centers in Spain. Eligible participants present FECD grade ≥2 on the modified Krachmer scale and have available preoperative Scheimpflug tomography and corneal densitometry measurements. The study population represents a real-world clinical cohort of patients routinely evaluated in corneal and cataract units, allowing assessment of the predictive performance and clinical utility of the SUCCESS Score under standard care conditions.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Need for endothelial keratoplasty (EK) after cataract surgery in patients with Fuchs endothelial corneal dystrophy | Up to 36 months after cataract surgery
  The primary outcome is the need for endothelial keratoplasty (EK) following phacoemulsification cataract surgery in patients with Fuchs endothelial corneal dystrophy (FECD). The endpoint is determined based on postoperative best-corrected visual acuity, corneal clarity, and presence of clinical signs of corneal decompensation. Each eye is evaluated using standardized follow-up visits and imaging criteria across participating centers. The decision to perform EK is made according to established clinical indications by the attending ophthalmologist, ensuring consistency across study sites.

SECONDARY OUTCOMES:
Model discrimination (Harrell's C statistic) of the SUCCESS Score | At primary analysis (October 2024)
  Model discrimination will be assessed using Harrell's C statistic (concordance index) to quantify how accurately the SUCCESS Score predicts the need for endothelial keratoplasty after cataract surgery in patients with FECD.
Calibration and predictive accuracy of the SUCCESS Score | At primary analysis (June 2026)
  Calibration plots and Brier score will be used to evaluate the agreement between predicted and observed probabilities of endothelial keratoplasty. Goodness-of-fit will be assessed across deciles of predicted risk.
Reclassification and clinical utility of the extended SUCCESS model | At primary analysis (June 2026)
  The incremental value of adding corneal densitometry to the SUCCESS Score will be assessed using Integrated Discrimination Improvement (IDI), Net Reclassification Improvement (NRI), and Decision Curve Analysis (DCA) to determine potential clinical benefit.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Ramón y Cajal, Universidad de Alcalá, Instituto Ramón y Cajal de Investigación Sanitaria (IRYCIS), Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data (IPD) that underlie the results reported in this article will be made available to qualified researchers upon reasonable request. Access will be granted after publication of the primary results and upon approval of a methodologically sound proposal. Data will be shared through a secure institutional platform of the Instituto Ramón y Cajal de Investigación Sanitaria (IRYCIS).
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning 12 months after publication and ending 36 months after publication.
Access Criteria: Qualified researchers affiliated with academic or non-profit institutions may request access to the deidentified individual participant data (IPD), study protocol, statistical analysis plan, and analytic code. Requests must include a methodologically sound proposal describing the intended analyses and objectives.
  Data and supporting materials will be shared through a secure institutional data repository managed by the Instituto Ramón y Cajal de Investigación Sanitaria (IRYCIS). Access will be granted upon approval by the study's data governance committee and completion of a data use agreement ensuring appropriate data handling and confidentiality.

REFERENCES:
- [Result] Arnalich-Montiel F, de-Arriba-Palomero P, Muriel A, Mingo-Botin D. A Risk Prediction Model for Endothelial Keratoplasty After Uncomplicated Cataract Surgery in Fuchs Endothelial Corneal Dystrophy. Am J Ophthalmol. 2021 Nov;231:70-78. doi: 10.1016/j.ajo.2021.04.016. Epub 2021 May 2. PMID 33951443